CLINICAL TRIAL: NCT00319917
Title: FK506 Phase 4 Study: A Double Blind Placebo Controlled Study to Assess the Efficacy on Joint Damage in RA Patients
Brief Title: A Double Blind Placebo Controlled Study to Assess the Efficacy on Joint Damage in RA Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-506-RA05
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Tacrolimus; Rheumatoid Arthritis; Tacrolimus anhydrous
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tacrolimus
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tacrolimus — oral
  Other Names: Prograf; FK506
  Arms: 1
Drug: placebo — oral
  Arms: 2

SUMMARY:
The purpose of the study is to assess the efficacy on joint damage and safety in RA patients treated with DMARDs in a double blind, placebo controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as rheumatoid arthritis by the revised ACR criteria
* Those who have been treated with an adequate stable dose of either methotrexate, salazosulfapyridine or bucillamine
* Those who have at least one erosion on X-ray of hands, wrists or feet

Exclusion Criteria:

* Those who have been treated with any biologic drugs or leflunomide
* Those who meet Class 4 with the Steinbrocker functional classification

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Radiographic progression of structural joint damage | 52 Weeks

SECONDARY OUTCOMES:
Signs and symptoms of rheumatoid arthritis | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chyugoku Region
  - Hokkaido Region
  - Hokuriku Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shin-etsu Region
  - Tohoku Region